CLINICAL TRIAL: NCT03376685
Title: The Relationship Between Exercise Frequency, Intensity, and Restoration of Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Jamie Burr, Dr. Jamie Burr, Director, Human Performance and Health Laboratory, Principal Investigator, Assistant Professor, PhD, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-08-008
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Overweight or Obesity
Keywords: Endurance training; Sprint interval training; Glycemic regulation; Lipid homeostasis; Cardiovascular health
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This study is a 6-week exercise training study, with two possible parallel training groups: endurance (END) or sprint (SIT) training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance Exercise Training (END) (Experimental): This group is performing END training for 6 weeks in duration. Intervention: Behavioral: Endurance Exercise Training (END)
  Interventions: Behavioral: Endurance Exercise Training (END)
- Sprint Exercise Training (SIT) (Experimental): This group is performing SIT training for 6 weeks in duration. Intervention: Behavioral: Sprint Exercise Training (SIT)
  Interventions: Behavioral: Sprint Exercise Training (SIT)

INTERVENTIONS:
Behavioral: Endurance Exercise Training (END) — Physical activity will be conducted on cycle ergometers under supervision. Participants will exercise 5 days a week for 30 minutes (Week 1-2); 35 minutes (Weeks 3-4); or 40 minutes (Weeks 5-6) at 60% VO2 peak.
  Arms: Endurance Exercise Training (END)
Behavioral: Sprint Exercise Training (SIT) — Physical activity will be conducted on cycle ergometers under supervision. Participants will exercise 3 days a week involving a 3-minute warm-up, followed up 4 repetitions (Week 1-2); 5 repetitions (Weeks 3-4); or 6 (Weeks 5-6) repetitions of 30 seconds at a maximal intensity with 2 minutes' rest in between. Exercise will conclude with a 2-minute cool-down.
  Arms: Sprint Exercise Training (SIT)

SUMMARY:
Regular physical activity is well established to decrease the risk of cardiometabolic diseases. While research has characterized responses based on exercise intensity, many beneficial effects of exercise are transient in nature, and therefore exercise frequency may play an important, yet currently under-appreciated, role in improving health. The purpose of this study is to determine the efficacy of 6-week high-frequency endurance (END) or low-frequency sprint (SIT) training with respect to reducing clinically relevant cardiometabolic risk factors in overweight/obese males. It is hypothesized that END, performed at a greater frequency than SIT, will markedly improve cardiometabolic health, while low-frequency SIT will not.

DETAILED DESCRIPTION:
Involvement in regular physical activity is known to elicit systemic adaptations and reduce the risk of cardiometabolic diseases, including hypertension, obesity, dyslipidemia, and hyperglycemia. Traditional physical activity recommendations suggest that 150 minutes of moderate-intensity continuous endurance (END) exercise dispersed over 5 days per week is sufficient to improve physical fitness in adults. However, given the commonly cited barrier of "lack of time," literature has recently focused on time effective sprint interval training (SIT), obtaining equivalent increases in aerobic capacity and acute glycemic regulation compared to classical END exercise when protocols are work-matched. Despite these similarities, END is conducive to daily sessions not feasible of SIT. As improvements in many clinically relevant risk factors are transient in nature following exercise, it remains imperative to assess the implications of variable frequency exercise regimes performed as per general practice (i.e. high-frequency END, low-frequency SIT). Furthermore, improvements in cardiovascular outcomes following END have been shown, in some instances, to be absent in response to SIT, suggesting END may be more beneficial for cardiovascular health. Therefore, the current study aims to assess several markers of cardiovascular (aerobic capacity, blood pressure, arterial stiffness, vascular endothelial function) and metabolic (glucose tolerance, lipid tolerance, body composition) health following 6-weeks of high-frequency END or low-frequency SIT, performed as per general practice. Combined, this research will provide important insight into the under-appreciated role of exercise frequency for improving cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-70 years
* Body mass index (BMI) > 25 kg/m^2 (classified as overweight or obese)
* Sedentary (<100 minutes moderate physical activity per week)
* Approval for vigorous exercise via physical activity readiness questionnaire (PARQ+)

Exclusion Criteria:

* Prescribed with glucose lowering medications
* Smoker
* Not cleared for physical activity

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via VO2 peak test, to determine the change in cardiorespiratory fitness following 6-weeks of exercise training
Free-living glycemic regulation | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via continuous glucose monitoring (CGM), to determine the change in free-living glycemic regulation following 6-weeks of exercise training
Glucose tolerance | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via an oral glucose tolerance test (OGTT) to determine changes in standardized glycemic regulation following 6-weeks of exercise training

SECONDARY OUTCOMES:
Blood lipids | Baseline (pre-training) vs. week 6 (post-training)
  Blood lipid profile from fasted venous blood sampling, including high-density lipoproteins (HDL), low-density lipoproteins (LDL), high-sensitivity C-reactive protein (Hs-CRP), cholesterol, non-HDL cholesterol, triglycerides (TAG), free-fatty acids (FFA), and cholesterol/HDL ratio
HbA1C | Baseline (pre-training) vs. week 6 (post-training)
  Change in HbA1C assessed via fasted venous blood sampling, following 6-weeks of exercise training
Post-prandial blood lipids | Baseline (pre-training) vs. week 6 (post-training)
  Assessed following the consumption of an oral fat tolerance test (OFTT). Blood lipid responses include triglycerides (TAG) and free fatty acids (FFA), assessing the influence of 6-weeks of exercise training on these parameters
Blood pressure | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via automated brachial blood pressure (including systolic (SBP), diastolic (DBP), and mean arterial pressure (MAP))
Body composition | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via dual-energy X-ray absorptiometry (DXA); including total and regional lean and fat mass. Assessed via height and weight measurements to determine BMI.
Arterial stiffness | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via carotid-femoral pulse wave velocity (PWV)
Arterial stiffness acutely post-exercise | Acutely pre-exercise vs. post-exercise in week 1 of training
  Assessed via carotid-femoral pulse wave velocity (PWV) following a single bout of exercise in week 1 of each group
Brachial artery vascular function | Baseline (pre-training) vs. week 6 (post-training)
  Assessed via brachial artery flow mediated dilation (FMD) following 6-weeks of exercise training
Brachial artery vascular function acutely post-exercise | Acutely pre-exercise vs. post-exercise in week 1 of training
  Assessed via brachial artery flow mediated dilation (FMD) following a single bout of exercise in week 1 of each training group
Daily sedentary/active time | Baseline (pre-training), week 1 (of training), week 6 (post-training)
  Assessed via accelerometer
Free-living glycemic regulation during the first week of exercise training | Baseline (pre-training) vs. week 1 (of training)
  Assessed via continuous glucose monitoring (CGM)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Burr, PhD, Principal Investigator — University of Guelph; Graham Holloway, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Petrick HL, King TJ, Pignanelli C, Vanderlinde TE, Cohen JN, Holloway GP, Burr JF. Endurance and Sprint Training Improve Glycemia and V O2peak but only Frequent Endurance Benefits Blood Pressure and Lipidemia. Med Sci Sports Exerc. 2021 Jun 1;53(6):1194-1205. doi: 10.1249/MSS.0000000000002582. PMID 33315809

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03376685/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03376685/SAP_003.pdf